CLINICAL TRIAL: NCT00623779
Title: A Controlled, Randomized, Parallel , Multi-centre Feasibility Study of the Oral Direct Thrombin Inhibitor, AZD0837, Given as ER Formulation, in the Prevention of Stroke and Systolic Embolic Events in Patients With Atrial Fibrillation, Who Are Appropriate for But Unable/Unwilling to Take VKA Therapy
Brief Title: Atrial Fibrillation (AF) Patients Not Taking Vitamin-K Antagonist (VKA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D1250C00051
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Results first posted 2011-07-28 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Persistent or Permanent Non-valvular Atrial Fibrillation
MeSH Terms: interventions — AZD 0837; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZD0837 — ER formulation
Drug: Aspirin — Oral form

SUMMARY:
The purpose of this study is to assess the safety and tolerability of AZD0837 in patients with atrial fibrillation who are unable or unwilling to take vitamin K antagonist therapy for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Either one of the following risk factors is sufficient for inclusion (high risk patient)
* Previous cerebral ischaemic attack (stroke or transient ischaemic attack (TIA), >30 days prior to randomization)
* Previous systemic embolism or at least one of the following risk factors are needed for inclusion: Age ≥75 years
* Symptomatic congestive heart failure
* Impaired left ventricular systolic function
* Diabetes mellitus; Hypertension requiring anti-hypertensive treatment
* In addition to AF the patient must be appropriate for but unable or unwilling to take VKA therapy

Exclusion Criteria:

* Presence of a clinically significant valvular heart disease;; Stroke or TIA and/or systemic embolism within the previous 30 days prior to randomization
* Conditions associated with increased risk of major bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Y Lip, MD, Principal Investigator — Birmingham City Hospital
Locations (38):
- Denmark (8):
  - Research Site, Aalborg
  - Research Site, Arhus N
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Frederikssund
  - Research Site, Horsens
  - Research Site, Silkeborg
  - Research Site, Svendborg
- Norway (6):
  - Research Site, Elverum
  - Research Site, Gjettum
  - Research Site, Kongsberg
  - Research Site, Oslo
  - Research Site, Stovner
  - Research Site, Straume
- Poland (13):
  - Research Site, Bytom
  - Research Site, Częstochowa
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Ostrów Mazowiecka
  - Research Site, Otwock
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Sopot
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Sweden (6):
  - Research Site, Borås
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Mölndal
  - Research Site, Stockholm
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Eastbourne
  - Research Site, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included male and female participants >18 years of age with chronic non-valvular Atrial Fibrillation. The participants were recruited during the time period from 22 October 2007 to 21 October 2008 at medical clinics in Europe.
Pre-assignment Details: For participants treated with Vitamin K Antagonists (VKA) at the time of enrollment, VKA treatment was to be adjusted (and stopped before randomisation) to ensure that INR was below 2.0 at randomisation. If this was not achieved the participant was discontinued from the study.
Groups:
- AZD0837 150 mg: AZD0837 150 mg
- AZD0837 300 mg: AZD0837 300 mg
- Standard Therapy: Standard Therapy
Period: Overall Study
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Started | 41 | 42 | 45
Completed | 38 | 39 | 44
Not Completed | 3 | 3 | 1
Not completed — Adverse Event | 1 | 3 | 0
Not completed — Criteria from CSR | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy | Total
Number analyzed (Participants) | 41 | 42 | 45 | 128
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.5 (8) | 71.6 (8.51) | 68.8 (9.36) | 70 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 17 | 49
  Male | 25 | 26 | 28 | 79

OUTCOME MEASURES:

1. Primary Outcome: Premature Discontinuation of Study or Study Drug Due to Any Reason
Description: The premature discontinuation of study or study drug due to any reason
Time Frame: 28 week (randomisation visit to last follow up visit in study) according to protocols
Measure: Number; unit: Participants
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 41 | 42 | 45
Participants | 4 | 6 | 3

2. Primary Outcome: Premature Discontinuation of Study Drug Due to Any Reason
Description: The premature discontinuation of study drug due to any reason
Time Frame: 24 weeks (randomisation visit to last treatment visit)
Measure: Number; unit: Participants
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 41 | 42 | 45
Participants | 3 | 3 | 1

3. Primary Outcome: Premature Discontinuation of Study Due to Any Reason
Description: |The premature discontinuation of study due to any reason
Time Frame: 28 weeks (randomisation visit to last follow up visit)
Measure: Number; unit: Participants
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 41 | 42 | 45
Participants | 4 | 4 | 2

4. Primary Outcome: Compliance With Study Drug
Description: [(number of doses dispensed-number of doses returned)/number of days between visits]*100
Time Frame: 24 weeks (randomisation visit to last treatment visit) according to protocol
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 41 | 39 | 0
Percentage | 96.95 (16.503) | 99.82 (11.383) |

5. Primary Outcome: Compliance With Study Visits/Assessments
Description: (number of visits attended acroos the time of study divided by the number of expected visits according to the time of entry into study)*100
Time Frame: 28 weeks (randomisation visit to last follow up visit) according to protocol
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 41 | 42 | 45
Percentage | 93.3 (15.01) | 95.6 (10.45) | 97.5 (6.8)

6. Secondary Outcome: Bleeding Events
Description: Number of patients with a bleeding event while on study drug. Patients with multiple bleeding events are counted once
Time Frame: 24 weeks (randomisation visit to last treatment visit) according to protocol. For patients who discontinued treatment the time frame was <24 weeks. Mean number of weeks was 7 weeks (baseline to end of treatment visit)
Population: 41 + 42 + 45 participants were randomized into the study to treatment arm 1, arm 2 and arm 3 respectively. However, one of the participants randomized to arm 2 was treated according to treatment arm 3
Measure: Number; unit: Participants
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 41 | 41 | 46
Participants | 0 | 5 | 2

7. Secondary Outcome: Change in Creatinine Level
Description: Individual change in Creatinine level (umil/L) from baseline to week 4 visit for patients while on study drug (week 4 visit-baseline)
Time Frame: 4 weeks according to protocol (randomisation visit to week 4 visit)
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 37 | 40 | 45
umol/L | 6.2 (8.64) | 3.6 (13.21) | 2.6 (12.90)

8. Secondary Outcome: Alanine Aminotransferase (ALAT)
Description: Number of patients while on study drug with Alanine aminotransferase (ALAT)>=3 times upper limit of normal.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 41 | 41 | 46
Participants | 0 | 0 | 1

9. Secondary Outcome: Bilirubin
Description: Number of patients while on study drug with Bilirubin>=2 times upper limit of normal.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 41 | 41 | 46
Participants | 1 | 0 | 0

10. Secondary Outcome: Plasma Concentration of AZD0837 (Prodrug)
Description: Assessment of plasma concentration of AZD0837 (prodrug) made on the week 4 visit
Time Frame: 4 weeks after baseline according to protocol
Measure: Median (Full Range); unit: nmol/L
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 24 | 26 | 0
nmol/L | 596.0 [5.0 to 2920.0] | 636.0 [18.2 to 5920.0] |

11. Secondary Outcome: Plasma Concentration of AR-H067637XX (Active Metabolite)
Description: Assessment of plasma concentration of AR-H067637XX (active metabolite) made on the week 4 visit
Time Frame: 4 weeks after baseline according to protocol
Measure: Median (Full Range); unit: nmol/L
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 24 | 26 | 0
nmol/L | 258.5 [5.0 to 539.0] | 368.5 [159.0 to 776.0] |

12. Secondary Outcome: Change in D-Dimer Level
Description: Individual change in D-Dimer level (ng/ml) from baseline to week 4 visit for patients while on study drug (week 4 visit-baseline)
Time Frame: 4 weeks according to protocol.(baseline to week 4 visit)
Measure: Median (Full Range); unit: ng/ml
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 38 | 38 | 43
ng/ml | -33.484 [-78.37 to 288.13] | -41.445 [-92.61 to 130.00] | 4.853 [-80.12 to 793.56]

13. Secondary Outcome: Activated Partial Thromboplastin Time (APTT)
Description: Individual change in Activated partial thromboplastin time (APTT) (sec) from baseline to week 4 visit for patients while on study drug (week 4 visit-baseline)
Time Frame: 4 weeks according to protocol.(baseline to week 4 visit)
Measure: Median (Full Range); unit: sec
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 25 | 20 | 0
sec | 31.74 [-17.8 to 105.8] | 51.51 [3.1 to 75.1] |

14. Secondary Outcome: Ecarin Clotting Time (ECT)
Description: Individual change in Ecarin clotting time (ECT) (sec) from baseline to week 4 visit for patients while on study drug (week 4 visit-baseline)
Time Frame: 4 weeks according to protocol.(baseline to week 4 visit)
Measure: Median (Full Range); unit: sec
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Number analyzed (Participants) | 24 | 18 | 0
sec | 125.6 [6 to 274] | 179.1 [7 to 341] |

ADVERSE EVENTS:
Description: 41 + 42 + 45 participants were randomized into the study to treatment arm 1, arm 2 and arm 3 respectively. However, one of the participants randomized to arm 2 was treated according to treatment arm 3
Arm/Group | AZD0837 150 mg | AZD0837 300 mg | Standard Therapy
Serious Adverse Events (participants affected / at risk) | 2/41 | 3/41 | 2/46
Other Adverse Events (participants affected / at risk) | 3/41 | 1/41 | 1/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0837 150 mg (N=41) | AZD0837 300 mg (N=41) | Standard Therapy (N=46)
Cardiac Failure (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Drug Intolerance (General disorders) | 0 | 1 | 0
Podagra (Metabolism and nutrition disorders) | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0837 150 mg (N=41) | AZD0837 300 mg (N=41) | Standard Therapy (N=46)
Bronchitis (Infections and infestations) | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less